CLINICAL TRIAL: NCT04538339
Title: Prediction of Arterial Lactate and Blood Gas Values Through the Analysis of Central Venous Blood. A Human, Prospective, Multicenter Validation Study.
Brief Title: Prediction of Arterial Lactate and Blood Gas Values Through the Analysis of Central Venous Blood
Acronym: PREDIGAZ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2020-11; 2020-A01333-36 (Other: IDRCB number issued by French Government)
Record Dates: First submitted 2020-08-29; First posted 2020-09-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Circulatory Failure
Keywords: Lactate; arterial blood gas; central venous blood; gazometer
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Predicting arterial lactate and blood gas values with sufficient accuracy by simply analyzing central venous blood would be interesting in intensive care unit patients in whom the insertion of an arterial catheter or arterial punctures could be avoided. This prospective study aims at externally validating published mathematical models built to predict arterial values from central venous blood analysis.

DETAILED DESCRIPTION:
Mathematical models for predicting arterial blood gas and arterial lactate have recently be published (PMID 27543529; see the citations section). The aim of the study is to externally validate these models in a multicenter (11 centres in France) cohort of intensive care unit patients suffering from acute circulatory failure. For the peru pose of the study, patients will undergo concomitent central venous/arterial blood sampling from 1 to 4 times during their intensive cafe unit stay. Clinical characteristics of the patients and central venous blood gas and lactate values will be used to predicted arterial values according to previously published formula. Predicted and actual arterial values of each variable of interest (pH, PaCO2, SaO2, lactate) will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* patient admitted in a intensive care unit
* patient already carrying an indwelling arterial catheter and a superior vena cava central catheter
* patient presenting an acute circulatory failure defined by the presence of at least two of the following items: a) Persistent hypotension (systolic arterial blood pressure < 90 mm Hg or mean arterial pressure < 65 mm Hg) or need for continuous intravenous vasopressor treatment (at any dose). b) Presence of at least one of the following signs of hypoperfusionfusion :Change in mental status ; Skin mottling ; Oliguria (Urine output <0.5 ml/kg body weight for at least one hour); Arterial lactate > 2 mmol/l or peripheral venous lactate > 3.2 mmol/l; ScvO2 <70%.
* Routine medical management requires central venous blood sampling for ScvO2 measurement and arterial blood sampling for gazometry.

Exclusion Criteria:

* Opposition to participation in the study
* Impossibility to take a concomitant arterial and venous gazometric sample.
* Patient treated with ECMO (extracorporeal membrane,oxygrnation), intermittent dialysis or continuous dialysis during sampling
* Patient hospitalized without consent and/or deprived of liberty by court decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Studied patients will be adult patients admitted to intensive car unit and presenting signs of acute circulatory failure. Patients should carry arterial and central venous catheters for their medical needs and not exclusively for the purpose of the study.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Percentage error rate when predicting arterial values (pH, PaCO2, SaO2 and lactate) from central venous values. | 15 minutes
  For each variable of interest (pH, PaCO2, SaO2 and lactate), the percentage of predicted values outside the agreement interval obtained in a previously published study (i.e., -0.078 to +0.084 for arterial pH; -1.32 to +1.36 kPa for PaCO2; -5.15 to +4.47% for SaO2; 1.07 to +1.05 mmol/l for arterial lactate) will be calculated.

SECONDARY OUTCOMES:
Bias and agreement interval between predicted and actual arterial values for each variable of interest. | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Toufik Kamel, MD, Principal Investigator — CHR Orléans, France
Locations (10):
- France (10):
  - CHU d'ANGERS, Angers
  - CHU de DIJON, Dijon
  - Chu de Garches, Garches
  - Chu Limoges, Limoges
  - Hopital de La Timone, Marseille
  - CHU de NANTES, Nantes
  - Chr D'Orleans, Orléans
  - CHRU de POITIERS, Poitiers
  - CHU de STRASBOURG, Strasbourg
  - Ch de Versailles, Versailles

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boulain T, Garot D, Vignon P, Lascarrou JB, Benzekri-Lefevre D, Dequin PF; Clinical Research in Intensive Care and Sepsis (CRICS) Group. Predicting arterial blood gas and lactate from central venous blood analysis in critically ill patients: a multicentre, prospective, diagnostic accuracy study. Br J Anaesth. 2016 Sep;117(3):341-9. doi: 10.1093/bja/aew261. PMID 27543529